CLINICAL TRIAL: NCT03498417
Title: Serum Antibodies Against the Insulin-like Growth Factor-1 Receptor (IGF-1R) in Graves' Disease and Graves' Orbitopathy
Brief Title: Anti-insulin-like Growth Factor-1 Receptor (IGF-1R) Antibodies in Graves' Disease and Graves' Orbitopathy
Acronym: IGF1RAbsGO
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Assistant Professor, University of Pisa
Other Study IDs: IGF1-R-Abs
Record Dates: First submitted 2018-03-30; First posted 2018-04-13 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Graves Ophthalmopathy; Graves Disease; Autoimmune Thyroiditis
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease; Thyroiditis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Graves' diseases: Patients with Graves' disease. No interventions foreseen
  Interventions: Diagnostic Test: Serum antibodies against the IGF-1R
- Autoimmune thyroiditis: Patients with autoimmune thyroiditis. No interventions foreseen
  Interventions: Diagnostic Test: Serum antibodies against the IGF-1R
- Healthy Subjects: Normal healthy subjects. No interventions foreseen
  Interventions: Diagnostic Test: Serum antibodies against the IGF-1R

INTERVENTIONS:
Diagnostic Test: Serum antibodies against the IGF-1R — Measurement of antibodies against the IGF-1R in serum samples by ELISA

SUMMARY:
The study is aimed at assessing IGF-1R-Abs in patients with Graves' disease, with or without GO, compared with healthy subjects and patients with autoimmune thyroiditis in a cross-sectional investigation.

ELIGIBILITY:
Inclusion Criteria:

1. for Graves' disease: a history of hyperthyroidism, associated with previous or present detectable serum autoantibodies against the TSH-R;
2. for autoimmune thyroiditis: the presence of at least two of the following: a) primary hypothyroidism; b) detectable serum autoantibodies against thyroglobulin or thyroperoxidase ; c) a hypoechoic pattern of the thyroid by ultrasound examination.
3. for healthy subjects: absence of any clinical, biochemical or instrumental evidence of thyroid diseases.

For all subjects: Informed consent

Exclusion Criteria:

1) lack of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with Graves' disease, with or without GO. The presence of GO will be established in any patient who had at least one of the following eye features: a) exophthalmometry ≥17 mm in women and ≥19 mm in men, based on measurements conducted for the normal population; b) eyelid aperture ≥9 mm; c) clinical activity score ≥1/7; iv) presence of diplopia; v) presence of corneal alterations; vi) presence of GO-related alterations of the fundi; and vii) reduction in visual acuity that could be attributed to GO.
  2. Patients with autoimmune thyroiditis
  3. healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Frequency of serum IGF-1R-Abs above the upper normal levels | Baseline
  Percent prevalence of serum IGF-1R-Abs above the upper normal levels in patients with GO, compared with healthy subjects, patients with Graves' disease without a clinically relevant GO, and patients with autoimmune thyroiditis.

SECONDARY OUTCOMES:
Serum concentrations of IGF-1R-Abs | Baseline
  Comparison of the serum concentrations of IGF-1R-Abs in patients with GO, compared with healthy subjects, patients with Graves' disease without GO, and patients with autoimmune thyroiditis;
Relationship between serum IGF-1R-Abs and the activity of GO | Baseline
  Relationship between serum IGF-1R-Abs (both levels and prevalence), with the the activity GO, namely the clinical activity score, including 7 items (spontaneous orbital pain, gaze provoked pain, palpebral redness, palpebral oedema, conjuctival redness, caruncle edema, chemosis) resulting in a score from 1 to 7
Relationship between serum IGF-1R-Abs and anti-TSH receptor autoantibodies | Baseline
  The relationship between serum IGF-1R-Abs (both levels and prevalence) and anti-thyrotropic hormone-receptor serum autoantibodies
Relationship between serum IGF-1R-Abs and anti-thyroperoxidase autoantibodies | Baseline
  The relationship between serum IGF-1R-Abs (both levels and prevalence) and anti-thyroperoxidase serum autoantibodies
Relationship between serum IGF-1R-Abs and anti-thyroglobulin autoantibodies | Baseline
  The relationship between serum IGF-1R-Abs (both levels and prevalence) and anti-thyroglobulin serum autoantibodies

CONTACTS AND LOCATIONS:
Overall Officials: Michele Marinò, MD, Principal Investigator — University of Pisa
Locations (1):
- Endocrinology Unit I, University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No